CLINICAL TRIAL: NCT06419166
Title: An Exploratory Clinical Study of GC012F Injection for the Treatment of Refractory Generalized Myasthenia Gravis
Brief Title: An Exploratory Clinical Study of GC012F Injection for Refractory gMG
Acronym: gMG
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The study stopped early, before enrolling its first participant.
Sponsor: Zhejiang University (Other)
Collaborators: Gracell Biotechnologies (Shanghai) Co., Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Director, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXB2024002
Record Dates: First submitted 2024-04-25; First posted 2024-05-17 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Refractory Generalized Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Refractory gMG subjects (Experimental): Refractory Generalized Myasthenia Gravis
  Interventions: Drug: GC012F injection

INTERVENTIONS:
Drug: GC012F injection — Each subject will receive GC012F injection (CD19-BCMA CAR-T cells) once by intravenous infusion on Day 0.
  Other Name: CD19-BCMA CAR-T cells

SUMMARY:
This study is a single-arm, open-label early exploratory clinical trial designed to evaluate the safety, tolerability, and preliminary efficacy of GC012F injection in subjects with refractory GMG. Additionally, the study aims to assess the pharmacokinetic (PK), pharmacodynamic (PD) characteristics, and immunogenicity of GC012F injection in subjects.

DETAILED DESCRIPTION:
This study is a single-arm, open-label early exploratory clinical trial designed to evaluate the safety, tolerability, and preliminary efficacy of GC012F injection in subjects with refractory GMG. Additionally, the study aims to assess the pharmacokinetic (PK), pharmacodynamic (PD) characteristics, and immunogenicity of GC012F injection in subjects.

The trial consists of several phases: screening period, apheresis day, baseline period, lymphodepletion period, pre-infusion assessment period, GC012F infusion period, safety and efficacy follow-up period, long-term follow-up period, and study discontinuation visit (if applicable).

Qualified subjects will undergo apheresis and receive the infusion after the production of CAR-T products. Subjects will undergo lymphodepletion before CAR-T cell infusion and assessment before infusion. Subjects meeting the cell infusion criteria will receive CAR-T cell infusion according to the dose specified in the protocol. Dose adjustments may occur based on safety and clinical efficacy for subjects in the same group or subsequent trial groups.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects or his/her legal proxy/guardian voluntary signing the ICF, and willing and able to follow the procedure in this study.
2. Aged ≥18 years old, no gender limitation;
3. Patients with confirmed refractory GMG, and the clinical classification is IIa-IVb (including IIa, IIb, IIIa, IIIb, IVa and IVb) in screening;
4. Patients whose MG-ADL score is 5 or more, and the proportion of ocular symptoms is less than 50% in the total score;
5. Patients with poor efficacy of conventional treatment and/or no effective treatment means relapse or exacerbation despite conventional hormone, immunosuppressant (e.g., azathioprine, mycophenolate mofetil, tacrolimus, cyclosporin A, cyclophosphamide, etc.), or rituximab treatment;
6. Patients who are on corticosteroids, the dose of prednisone should not exceed 20 mg/d (or no more than an equivalent dose of another corticosteroid) during the 3 weeks prior to apheresis, and the dose isn't escalated during 3weeksk prior to apheresis, the dose isn't changed within 4 weeks prior to infusion;
7. Patients with positive MG-specific autoantibodies in the screening period: acetylcholine receptor autoantibody (anti-AChR) titer or muscle-specific tyrosine kinase autoantibody (anti-MuSK) or low-density lipoprotein receptor-associated protein 4 autoantibody (anti-LRP4) or anti-acetylcholine receptor cluster antibody must be higher than the upper limit of the laboratory reference normal value;
8. Life expectancy ≥3 months;
9. The results of laboratory test during screening period shall meet all following criteria:

   1. Neu ≥1.0 × 109/L; Hb ≥8.0 g/dL; PLT ≥50 × 109/L;
   2. ALT ≤3 × ULN; AST ≤3 × ULN; TBIL <2 × ULN (DBIL ≤1.5 × ULN for subjects with Gilbert's syndrome)
   3. Creatinine clearance (19.3 Appendix 3) ≥30 mL/min;
   4. APTT ≤1.5 × ULN, PT ≤1.5 × ULN;
   5. LVEF ≥50% based on echocardiography, no findings of pericardial effusion.
10. Women of child-bearing age should:

    1. Have a negative serum β human chorionic gonadotropin (β-hCG) pregnancy test confirmed by investigators during the screening period;
    2. Agree to avoid breastfeeding during the study period until at least 1 year after the infusion of GC012F Injection or until two consecutive flow cytometry tests show the absence of CAR-T cells (whichever occurs later).
11. Any male subjects who have sexual partners and female subjects with childbearing potential shall agree to take effective contraceptive methods (e.g. oral contraceptive pills, intrauterine device or condoms) from the screening starting until at least 1 year post GC012F Injection infusion or until two consecutive flow cytometry tests show the absence of CAR-T cells (whichever occurs later. Male subjects must agree to use condoms during sexual contact with pregnant females or females with fertility for at least 1 year after the infusion of GC012F Injection, even if a successful vasectomy has been performed;
12. Venous access available for blood collection, and no contraindications for leukapheresis.

exclusion criteria:

1. Subjects have a history of severe hypersensitivity or allergy;
2. Any contraindication for fludarabine, cyclophosphamide and any component of the investigational product;
3. Subjects with any of the following heart diseases:

   1. Congestive heart failure (New York Heart Association (NYHA) Class III or IV);
   2. Experienced myocardial infarction or underwent coronary artery bypass grafting (CABG) within 6 months prior to screening period;
   3. Clinically significant ventricular arrhythmias or a history of unexplained syncope not due to vasovagal reaction or dehydration; or a QTc interval >480 ms during screening;
   4. History of severe non-ischemic cardiomyopathy.
4. Accompanied by other uncontrolled malignancies. Subjects with the following conditions should be excluded: early-stage tumors that have received radical treatment (carcinoma in situ or grade 1 tumors, or non-ulcerated primary melanoma with a depth <1 mm and no involvement of lymph nodes), basal cell skin cancer, skin squamous cell carcinoma, cervical carcinoma in situ, or breast cancer in situ that has received potential radical treatment;
5. Severe underlying medical conditions, such as:

   1. Fungal, bacterial, viral or other infections or suspected fungal, bacterial, viral or other infections that cannot be controlled or require general intravenous administration;
   2. Significant clinical evidence of dementia or mental status changes;
   3. History of any central nervous system (CNS) or neurodegenerative diseases, (e.g., epilepsy, seizures, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, psychiatric disorders).
6. Positive results in any of the following tests:

   1. HIV antibody positive;
   2. HBsAg positive; or HBcAb positive and HBV-DNA above the lower limit of detection of the analytical method;
   3. HCV antibody positive with HCV RNA above the lower limit of detection of the analysis method; or known history of hepatitis C without completion of antiviral therapy for ≥24 weeks;
   4. Syphilis antibody positive.
7. Received therapy of non-hormonal immunosuppressants within 3 weeks prior to apheresis;
8. Major surgery within 2 weeks prior to leukapheresis or surgery plan during the study (except for local anesthesia surgery, but not performed within 2 weeks after infusion);
9. Receipt of a live-attenuated vaccine within 4 weeks prior to leukapheresis;
10. Intravenous injection of immunoglobulins or therapy of plasma exchange (PE);
11. Receipt of other biologics for MG within 3 weeks prior to apheresis or within 8 weeks prior to infusion;
12. Participation in any other clinical trial within 4 weeks prior to signing ICF, or the date of signing the ICF still within 5 half-lives of the drug from the last dose in the last clinical trial (whichever is longer);
13. Thymectomy within 12 months prior to ICF signing;
14. Pregnant women or lactating women who do not agree to abstain from breastfeeding, men and women who have a fertility plan during participation in this study or within 1 year after receiving study treatment;
15. Any situation that may hinder subjects' participation in the entire trial or confuse the results, or any situation in which investigators believe that participation in this study is not in the subject's best interests.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLT | Within 28 days after GC012F injection infusion
  DLT
Frequency and severity of abnormal findings in electrocardiograms | Within 96 weeks after GC012F injection infusion
  The electrocardiography shall be measured after 5 minutes of rest, and assessments included as follows: Heart rate, RR interval, PR interval, QT interval, QRS wave, QT interval and other indexes.
Frequency and severity of abnormal findings of adverse events. | Within 96 weeks after GC012F injection infusion
  Any untoward medical event that occurs after a subject has administered an investigational product, which may be manifested as a symptom, sign, disease or laboratory abnormality but does not necessarily have a causal relationship with the investigational product.
Frequency and severity of abnormal findings in physical examinations | Within 96 weeks after GC012F injection infusion
  The full physical examination at least includes assessments of skin, mucosa, lymph nodes, head, neck, chest, abdomen, spine/limbs, and nervous system. A full physical examination needs to be completed only during the screening period, and the physical examination can be performed in subsequent visit as per changes in signs and symptoms.
Frequency and severity of abnormal findings in laboratory tests | Within 96 weeks after GC012F injection infusion
  Laboratory tests include blood test，Coagulation function ，Infectious disease detection and tests recommended by the Investigator
Frequency and severity of abnormal findings in vital signs | Within 96 weeks after GC012F injection infusion
  Vital signs shall be measured after 5 minutes of rest, and assessments included as follows: Temperature, oxygen saturation, heart rate, respiratory rate, resting systolic and diastolic blood pressure.
RP1D | 2 years after GC012F injection infusion
  Recommended phase I dose
MTD | 2 years after GC012F injection infusion
  maximum tolerated dose

SECONDARY OUTCOMES:
PK parameters of CAR-T cells in peripheral blood after GC012F infusion (Cmax); | Within 96 weeks after GC012F injection infusion
  PK results of GC012F
PK parameters of CAR-T cells in peripheral blood after GC012F infusion (Tmax); | Within 96 weeks after GC012F injection infusion
  PK results of GC012F
PK parameters of CAR-T cells in peripheral blood after GC012F infusion ( AUC); | Within 96 weeks after GC012F injection infusion
  PK results of GC012F
Levels of cytokines [IL-6、IL-10、IFN-γ、TNF-α、MCP-1(as applicable)], lymphocyte subsets, and soluble BCMA in peripheral blood after GC012F infusion; | Within 28 days after GC012F injection infusion
  PK results of GC012F
Disease activity indices:MG-ADL | Within 96 weeks after GC012F injection infusion
  Efficacy results of GC012F
Disease activity indices:MGC | Within 96 weeks after GC012F injection infusion
  Efficacy results of GC012F
Disease activity indices:QMG | Within 96 weeks after GC012F injection infusion
  Efficacy results of GC012F
Disease activity indices: MG-QoL 15r | Within 96 weeks after GC012F injection infusion
  Efficacy results of GC012F
Disease activity indices: post-intervention status according to the Myasthenia Gravis Foundation of America (MGFA) classification | Within 96 weeks after GC012F injection infusion
  Efficacy results of GC012F

OTHER OUTCOMES:
• Detection rate of CAR-T cell antibodies in peripheral blood within 24 weeks post-GC012F infusion; | within 24 weeks post-GC012F infusion;
  Safety of GC012F
• Changes in serum immunoglobulin levels (including IgG, IgM, IgA, and IgE) in patients within 24 weeks post-GC012F infusion; | within 24 weeks post-GC012F infusion
  Safety of GC012F
• Detection rate of replication-competent lentivirus (RCL). | Within 15 years after GC012F injection infusion
  Safety of GC012F

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital,College of Medicine, Zhejiang University, Hanzhou, Zhejiang, China